CLINICAL TRIAL: NCT03686189
Title: Safety and Efficacy Study of Iliac Bifurcation Stent Graft System, A Prospective, Multi-centre, Single-Arm Clinical Trial
Brief Title: Safety and Efficacy Study of Iliac Bifurcation Stent Graft System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50CT（CN）
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Aortoiliac Aneurysm; Iliac Aneurysm
Keywords: Iliac Bifurcation Stent Graft System
MeSH Terms: conditions — Iliac Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Participants will be treated with Iliac Bifurcation Stent Graft System
  Interventions: Device: Iliac Bifurcation Stent Graft System

INTERVENTIONS:
Device: Iliac Bifurcation Stent Graft System — Device placement after preoperative preparation. For patients with the aortoiliac aneurysm, the placement of short-bodied iliac artery bifurcation stent graft combined with the placement of the abdominal aortic stent graft, or the placement of long-bodied iliac artery bifurcation stent graft combined with the placement of the abdominal aortic stent graft are recommended.

SUMMARY:
A prospective, multi-centre, single-arm clinical trial to evaluate the safety and efficacy of Iliac Bifurcation Stent Graft System.

DETAILED DESCRIPTION:
A prospective, multi-center, Single-Arm clinical trial to evaluate the safety and efficacy of endovascular treatment of the aortoiliac aneurysm or the iliac aneurysm by using Iliac Bifurcation Stent Graft System manufactured by Lifetech Scientific (Shenzhen) Co., LTD. According to the requirements of the study, 64 patients preoperatively diagnosed with the aortoiliac aneurysm or the iliac aneurysm will be recruited and be treated by Iliac Bifurcation Stent Graft System under the guidance of aortic aortography. The safety of operations, stability of releasing stent and the accuracy of positioning will be evaluated intraoperatively. The safety and efficacy of aortic endovascular treatment of Iliac Bifurcation Stent Graft System will be observed by postoperative follow up scheduled 30 days and 180 days after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years of age.
2. The subject or its legal representative sign the informed consent.
3. Patients with the aortoiliac aneurysm or the iliac aneurysm and need to endovascular restructure the internal iliac artery.
4. The anatomical structure of the iliac artery meets the following requirements:

   1. The length of the anchoring zone of the external iliac artery is ≥15mm.
   2. The diameter of the anchoring zone of the external iliac artery is between 7mm and 12mm.
   3. The diameter of the external iliac artery is between 6mm-10mm.
   4. The length of the anchoring zone of the internal iliac artery is ≥10mm.
5. Life expectancy is longer than one year.

Exclusion Criteria:

1. The patient is under 18 years old.
2. Pregnant or lactating woman.
3. The patient had a myocardial infarction or stroke within 3 months.
4. The patient had connective tissue disease, infectious aneurysm, and other active infections.
5. The patient has abdominal aortic aneurysm rupture.
6. The patient has a severe coagulation disorder.
7. Allergic to the material of stent or contrast media.
8. Patient's vascular morphology is not suitable for endovascular repairs, such as serious stricture, dilate, bend, sclerosis, etc. of the iliac artery.
9. Patients with severe mural thrombus in the aneurysm cavity, which may affect the implantation of Branch Stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Patency rate of internal iliac artery | 180days postoperative
  Patency rate of internal iliac artery >＝89%

SECONDARY OUTCOMES:
Technical success rate | immediate
  After implantation of the stent and observed under common iliac artery angiography, the stent was in the right position and adhered well to the vessel wall, with no leakage.
Clinical success rate | 30 days and 180days postoperative.
  The diameter of the common iliac artery aneurysm was not expanded or expanded less than 3mm.
The incidence of major Adverse Device Effects (ADEs) | Before discharge, 30 days and 180 days postoperative。
  Major Adverse Device Effects including death, myocardial infarction, arterial thrombosis, renal function failure, respiratory failure, paraplegia, stroke, gluteus claudication, colon, spinal cord ischemia necrosis, perineum, iliac artery blockages, external iliac vein blockage, expand common iliac artery aneurysms (increased diameter 3 mm), common iliac artery aneurysms rupture, internal leakage (type I and type III), stent fracture, stent displacement.
Device related mortality | Before discharge, 30 days and 180days postoperative.
  Deaths related to the device.
Secondary interventional surgery | Before discharge, 30 days and 180days postoperative.
  The rate of secondary interventional surgery for complications related to the device

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Principal Investigator — Chinese PLA General Hospital
Locations (8):
- China (8):
  - Beijing Anzhen Hospital, Capital Medical university, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Frist Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Jiangsu Province Hospital, Nanjing